CLINICAL TRIAL: NCT03708055
Title: Prevention of Frailty in Breast Cancer Survivors: A Pilot Study
Brief Title: Weight Bearing Exercise in Preventing Frailty in Stage I-IIIA Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0800000618; NCI-2018-01888 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0800000618 (Other: The University of Arizona); P30CA023074 (NIH)
Record Dates: First submitted 2018-10-09; First posted 2018-10-16 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Cancer Survivor; Overweight; Postmenopausal; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (weight bearing exercise program) (Experimental): Participants undergo a weight bearing exercise program in a group 2 days a week and at home 5 days a week for 8 weeks.
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — Undergo weight bearing exercise program

SUMMARY:
This trial studies how well weight bearing exercise works in preventing frailty in stage I-IIIA breast cancer survivors. Weight bearing exercise, including muscle-strengthening, aerobic, flexibility, and balance exercises, can decrease fat and increase muscle, which may lead to reduced frailty.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate reproducibility of forearm muscle activation and subcutaneous fat measures in a healthy convenience sample/population (N= 10).

II. Demonstrate that measures of muscle activation and signal attenuation by subcutaneous fat mass can be conducted in a systematic and reproducible fashion in breast cancer survivors prior to and following weight bearing exercise training.

III. In a cross sectional analysis, describe the level of lean muscle mass, muscle activation, strength, insulin resistance, inflammatory cytokines and growth factors, and inter-individual variability in breast cancer survivors prior to training.

IV. Describe the level of lean muscle mass, muscle activation, strength, insulin resistance, inflammatory cytokines (such as IL-6, CRP and others), and growth factors (such as myostatin, IGF-1, IGFBP-3 and others) in breast cancer survivors following weight bearing exercise training.

V. Evaluate the influence of genetic variability on response to prescribed training in breast cancer survivors.

OUTLINE:

Participants undergo a weight bearing exercise program in a group 2 days a week and at home 5 days a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal (12 months without menstrual period: naturally, surgically, by hormone suppression).
* History of early stage breast cancer (stage I, II, IIIa).
* At least 6 months from chemotherapy.
* May be receiving hormonal therapy during the study.
* Currently disease-free, including a negative mammogram within 1 year.
* Body mass index (BMI) between 25 and 40kg/m^2.
* In general good health with no acute or chronic disease that could worsen with weight bearing exercise.
* Not currently on a prescribed diet nor reporting weight loss of > 10 pounds (lbs) in previous 3 months.
* Not currently participating in physical activity (PA) independently or a structured program (performing < 120 min of low-intensity, low-impact exercise per week; and no weightlifting or similar physical activity).
* Ability to participate in physical activity, not limited by severe disability (e.g., severe arthritic conditions); chronic back pain, or history or presence of diseases for which increased physical activity would not be advised.
* No severe chronic disease, other than breast cancer (e.g., human immunodeficiency virus/acquired immunodeficiency syndrome [HIV/AIDS], kidney failure, liver failure, chronic obstructive pulmonary disease, congestive heart failure, Alzheimer?s, unstable angina, uncontrolled asthma, uncontrolled diabetes, uncontrolled hypertension).
* No implanted cardiac pacemaker, cardiac defibrillator, or other implanted electronic medical equipment.
* No history of drug or alcohol abuse.
* Able to remain in a lying or sitting position for an extended period (> 30 minutes).
* No history or presence of a significant psychiatric disorder or any other condition that would interfere with participation in the trial.
* Medical clearance by treating physician.
* Willing to discontinue nonsteroidal antiinflammatory drug (NSAID) use, except Tylenol and baby aspirin (80mg), 1 week prior to blood draws.
* Willing to maintain body weight during the study.
* Can be reached by telephone.
* Willing to complete consent process and sign informed consent form.

Ages: 37 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-07-24 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Reproducibility of muscle activation by subcutaneous fat mass measures. | Up to 9 years
  Demonstrate reproducibility of forearm muscle activation and subcutaneous fat measures in a healthy convenience sample/population (N= 10). Standard anthropometric measurements (height, weight, waist, hip and arm circumferences) will be taken at baseline and 8weeks. A total body dual energy X-ray absorptiometry (DXA) scan, with an effective radiation dose of about 0.01 mSv, which is about the same as background radiation in one day according to the American College of Radiology (http://www.radiologyinfo.org/en/safety/index.cfm?pg=sfty_xray#3), will be used to determine fat mass and fat free mass at these same time-points. Skeletal muscle mass will be determined by using both appendicular lean mass/height2 method and the residuals model from the Health ABC Study.
Amount of lean muscle as determined by using both appendicular lean mass/height2 method and the residuals model from the Health ABC Study. | 8 weeks
  Skeletal muscle mass will be determined by using both appendicular lean mass/height2 method and the residuals model from the Health ABC Study.
Reproducibility of signal attenuation using electromyography (EMG) | Up two weeks
  Maximal isometric muscle activation of the forearm flexors by electromyography (EMG) will be assessed by a pair of surface electrodes (plus 1 ground), to minimize participant burden. EMG data will be amplified and recorded by BIOPAC Systems MP35, 4-channel acquisition system and BSL Pro 3.7 software (BIOPAC Systems, Inc. Goleta, CA), during each of 4, 2-second, repetitions on the 100kg hand grip isometric dynamometer, integrated into the BIOPAC system. Sampling rate and acquisition length will be standardized. The I-beam tool will select the initiation of and conclusion of each contraction. Contraction 1 for each participant will be used for exercise familiarization and dropped, contractions 2-4 will be averaged to for maximal isometric muscle activation (mV). Normally, the non-dominant arm would be evaluated, but since this particular population may have functional limitations on either or both sides due to surgery (i.e. lymphectomy or mastectomy), both arms will be measured.
Level of strength as measured by 8-12 repetition maximum (RM) and by hand grip dynamometer. | Up to 8 weeks
  A standard submaximal test of strength, 8-12 repetition maximum (RM) will used to evaluate strength and maintain loads in the lower body, which has been safe and effective in previous studies. Strength by hand grip dynamometer will also be measured at baseline and 8wks post-training.

OTHER OUTCOMES:
Measure changes in biomarkers, i.e. insulin resistance, inflammatory cytokines (such as IL-6, CRP and others), and growth factors (such as myostatin, IGF-1, IGFBP-3 and others). | Up to 8 weeks
  Insulin, insulin resistance (homeostasis model of insulin resistance, HOMA-IR), growth factors and pro-inflammatory cytokines will be evaluated. Assays will be performed in duplicate for insulin and in triplicate for glucose, based on prior assay experience, with baseline and 8 wk samples for each individual run within the same assay. An Insulin Radioimmunoassay Kit will be used to quantify fasting insulin levels.Determination of glucose will be performed by colorimetric assay via the glucose oxidase method and spectrophotometer. Past intra- and inter-assay CVs were 5% and 8% for glucose measures respectively. HOMA-IR = insulin0 (uU/ml)*glucose0 (mmol/l)) / 22.5.
  Highly sensitive ELISA kits will be used to measure circulating cytokines, such as IL-6 or CRP and growth factors, such as IGF-1 in duplicate. Controls for each assay will be run concurrently on each plate. Each assay will be run with intra and inter assay CVs of <5% and <10% respectively.
Quantitative and qualitative analysis of DNA. | Up to 8 weeks
  DNA extraction from blood buffy coat or whole blood will be performed using the FlexiGene DNA Kit following the protocol for Isolation of DNA from 100-500µl Buffy Coat. Quantitative and qualitative DNA analysis will be performed by the Quant-iT™ PicoGreen® dsDNA Assay Kit and by performing 558bp polymerase chain reaction (PCR) and separation by gel electrophoresis on a 2% agarose gel, stained with ethidium bromide for visualization. Determination of polymorphisms related to body composition, exercise or chronic disease will be performed using TaqMan® Pre-Designed SNP Genotyping Assays with allelic discrimination by the ABI PRISMTM 7700 Sequence Detector. If TaqMan technology is not suitable for a particular polymorphism, then simple multiplex PCR with primers designed by Midland Chemicals will be performed and allelic determination will be conducted by ethidium bromide visualization on agarose gel. Universal PCR thermocycling conditions will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Bea, Principal Investigator — The University of Arizona Medical Center-University Campus
Locations (1):
- The University of Arizona Medical Center-University Campus, Tucson, Arizona, United States